CLINICAL TRIAL: NCT00684008
Title: A Phase I Study of CYT107 (Recombinant Glycosylated Human IL-7) in Recipients of HLA Matched Ex Vivo T Cell Depleted Bone Marrow or Peripheral Blood Stem Cell Transplant
Brief Title: Safety Study of IL-7 in Recipients of a Hemopoietic Stem Cell Transplant Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytheris, Inc. (Industry)
Responsible Party: Marcel R.M. van den Brink, M.D., Ph.D., Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-08; MSKCC IRB #07-127
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: AML; CML; MDS
Keywords: interleukin-7; immune based therapies; graft vs host disease; immune reconstitution; infection; lymphopenia; hematopoetic stem cell transplantation; bone marrow transplantation; peripheral blood stem cell transplant; immunosuppression
MeSH Terms: conditions — Graft vs Host Disease; Infections; Lymphopenia | interventions — efineptakin alfa; Interleukin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Single arm dose escalation study. Three successive cohorts of 3 patients each. Doses to be evaluated: 10, 20, and 30 mcg/kg/dose for 3 consecutive doses.
  CYT107 is a recombinant protein belonging to the class of growth factors known as cytokines.
  CYT107 is a heavily glycosylated and sialylated form of recombinant human Interleukin-7.
  CYT107 is supplied as a sterile colorless liquid at a concentration of 4 mg/ml.
  Interventions: Drug: CYT107 - Recombinant glycosylated human interleukin 7.; Drug: rhIL-7 (CYT107)

INTERVENTIONS:
Drug: CYT107 - Recombinant glycosylated human interleukin 7. — Patients will be treated with CYT107 60 to 210 days post transplantation, in 3 successive cohorts of 3 patients. Escalating doses of CYT107 will be given to successive cohorts. Patients will receive 1 dose of CYT107 by the subcutaneous route, once a week for 3 weeks. Dose level 1: 10 mcg/kg/dose for 3 doses; Dose level II: 20 mcg/kg/dose for 3 doses; Dose level III: 30 mcg/kg/dose for 3 doses. Only 1 treatment course for this initial study.
  Other Names: rhIL-7
Drug: rhIL-7 (CYT107) — 10, 20, or 30 mcg/kg once a week for 3 consecutive weeks via the subcutaneous route.
  Other Names: interleukin-7

SUMMARY:
This is a phase I inter-patient dose escalation open labeled study assessing multiple doses of CYT107 in patients of at least 15 years of age, who are recipients of HLA matched ex vivo T cell depleted bone marrow or peripheral blood stem transplants.

The dose escalation design is aimed at establishing the absence of significant toxicity and to define a biologically active dose in this patient population.

At each dose level, eligible patients will receive 3 doses of CYT107 injected subcutaneously (under the skin of the arm, legs, or stomach) once a week for 3 weeks.

Groups of three patients will be entered at each dose level of CYT107. Three dose levels are planned: 10 mcg/kg/week, 20 mcg/kg/week and 30 mcg/kg/week. Three patients must complete day 42 of the study at a dose level without a dose limiting toxicity (DLT) before there is escalation to the next dose level.

DETAILED DESCRIPTION:
Rationale: Delayed and deficient reconstitution of T cells and their functions are a major obstacle to the success of a hematopoietic stem cell transplant (HSCT). CYT-107 may have potential clinical use after allogeneic HSCT to enhance lymphoid reconstitution which could have a number of beneficial effects including decreased morbidity and mortality from post-transplant infections. Our preliminary data with a previous generation IL-7, CYT 99 007, raise the possibility that IL-7 could have, in some cases, an anti-GVHD effect while keeping the anti-tumor effect of the allograft intact.

Primary Objective:

* To determine the safety and a recommended dose of CYT107 (r-hIL-7) in recipients of an HLA-matched related or unrelated ex vivo T-cell-depleted bone marrow (BM) or peripheral blood stem cell (PBSC) transplant after initial engraftment and hematopoietic reconstitution.
* If toxicities are encountered, to establish the maximum tolerated dose (MTD) and dose limiting toxicities (DLT).

Secondary Objectives:

* To define the pharmacokinetics of escalating doses of CYT107 in recipients of allogeneic transplants.

To achieve preliminary characterization:

* Of the effects of CYT107 treatment on engraftment and GVHD.
* Of the effects of CYT107 on the recovery of T, NK and B cell populations and their functions in vitro.
* Of a tolerable biologically active range of doses for CYT107 in recipients of allogeneic transplants.
* Whether and to what degree administration of CYT107 might influence the risk of developing an EBV-lymphoproliferative disorder.
* Of the effects of CYT107 treatment on leukemia relapse.

ELIGIBILITY:
Inclusion Criteria:

* Able to read consent form and give informed consent.
* At least 15 years old.
* Histologically confirmed non-lymphoid hematological malignancy.
* Recipient of T cell depleted bone marrow (BM) or peripheral blood stem cell (PBSC) transplant from a 6/6 HLA (A, B, DR by intermediate resolution) identical related or unrelated donor after myeloablative conditioning.
* Received TCD HCT containing < 1x105 CD3+ T cells/kg of recipient.
* Patient included in at least one of the following categories:

  * AML in 2nd or greater complete remission.
  * High-risk AML (high-risk cytogenetics, undifferentiated leukemia, secondary AML, antecedent MDS) in 1st remission.
  * CML in 2nd or greater chronic phase, 2nd or greater accelerated phase.
  * MDS intermediate or high risk by IPSS criteria.
* History of opportunistic infection (CMV viremia requiring anti-viral therapy, PCP pneumonia, mycobacterial infection, herpes zoster, viral respiratory infection (influenza, RSV, para-influenza), etc.
* CD4+ T cell count < 100 at 6 months post-transplant.
* At high risk for opportunistic infection (e.g., history of treated invasive fungal infection prior to the transplantation, positive CMV serology in patient, or positive toxoplasmosis serology in donor and patient, etc.).
* 60 - 210 days post transplant.
* In remission at the time of initiation of CYT107.
* Documented engraftment with sustained neutrophil counts of at least 1000/mcl and untransfused platelet counts > 20 000/mcl for 3 consecutive lab values (the last one tested <10 days before initiation of treatment) on 3 different days prior to treatment. Patients who have engrafted but require G-CSF for myelosuppressive antibiotics or antiviral medications are eligible if they require G-CSF no more than twice weekly and their ANC remains >1000/mcl.
* KPS > 60%.
* Adequate organ function:

  * Cardiac: No evidence of change in cardiac function by history, exam and/or EKG post-HCT.
  * Pulmonary: Absence of dyspnea or hypoxia (< 90% of saturation by pulse oxymetry on room air).
  * Hepatic: Bilirubin <= 1.5 X ULN, AST (SGOT) and /or ALT (SGPT) <= 2.5 X ULN. PT/PTT < 1.5 X ULN.
  * Renal: Calculated Creatinine clearance > 60 mL/min/1.73 m2. [Note: all transplant patients had an ejection fraction of > 40% on their pre-transplant echocardiogram and a DLCO > 50% of predicted (corrected for hemoglobin)]

Exclusion Criteria:

* No evidence or history of acute GVHD or of chronic GVHD.
* No recurrent leukemia post HCT.
* No active uncontrolled viral, bacterial or fungal infection.
* No documented HIV-1 or -2, HBV or HCV infection at any time before or after transplant (a positive hepatitis B serology indicative of a previous immunization is not an exclusion criteria).
* Not be receiving systemic corticosteroid, anti-mitotic agent or other immunosuppressive treatment.
* Not receiving Growth Hormone or gonadotropin agonists/ antagonists.
* Not receiving any cytokine support other than G-CSF post-HCT.
* Not receiving concurrent treatment with another investigational drug and/or biological agent.
* Not receiving anticoagulant therapy.
* No uncontrolled hypertension.
* No history of lymphoid malignancy (e.g. Hodgkin disease, non Hodgkin lymphoma, Acute Lymphoblastic Leukemia and Chronic Lymphocytic Leukemia) or acute biphenotypic leukemia.
* No peripheral lymphadenopathy (any lymph node > 1 cm).
* No history of EBV associated lymphoproliferation.
* No EBV viremia equal to or greater than 500 copies EBV DNA/mL of blood by quantitative PCR.
* No history of autoimmune disease nor a HCT donor with a history of an autoimmune disease.
* Fertile patients must use effective birth control. Not pregnant or nursing. Negative pregnancy test within 2 weeks of study treatment.
* QTc prolongation (QTc > 470 ms) or prior history of significant arrhythmia or ECG abnormalities.
* No active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Any past or current psychiatric illness that, in the opinion of the investigator, would interfere with adherence to study requirements or the ability and willingness to give written informed consent.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Toxicity of CYT107 in post-transplant patients with AML, CML and MDS using the NCI Common Toxicity Criteria version 3.0 with the BMT specific adverse event grading system. | Visits: 2 week screening period; treatment visits on days 0, 7, and 14; non-treatment visits on Days 1, 21, 28, 42, 56, and 77.

SECONDARY OUTCOMES:
Pharmacokinetics and Pharmacodynamics | Study days 0, 1, 7, 14, 21, 28, 42, and 77.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel van den Brink, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Institute, New York, New York, United States

REFERENCES:
- [Background] Alpdogan O, Muriglan SJ, Eng JM, Willis LM, Greenberg AS, Kappel BJ, van den Brink MR. IL-7 enhances peripheral T cell reconstitution after allogeneic hematopoietic stem cell transplantation. J Clin Invest. 2003 Oct;112(7):1095-107. doi: 10.1172/JCI17865. PMID 14523046
- [Background] Rosenberg SA, Sportes C, Ahmadzadeh M, Fry TJ, Ngo LT, Schwarz SL, Stetler-Stevenson M, Morton KE, Mavroukakis SA, Morre M, Buffet R, Mackall CL, Gress RE. IL-7 administration to humans leads to expansion of CD8+ and CD4+ cells but a relative decrease of CD4+ T-regulatory cells. J Immunother. 2006 May-Jun;29(3):313-9. doi: 10.1097/01.cji.0000210386.55951.c2. PMID 16699374
- [Derived] Perales MA, Goldberg JD, Yuan J, Koehne G, Lechner L, Papadopoulos EB, Young JW, Jakubowski AA, Zaidi B, Gallardo H, Liu C, Rasalan T, Wolchok JD, Croughs T, Morre M, Devlin SM, van den Brink MR. Recombinant human interleukin-7 (CYT107) promotes T-cell recovery after allogeneic stem cell transplantation. Blood. 2012 Dec 6;120(24):4882-91. doi: 10.1182/blood-2012-06-437236. Epub 2012 Sep 25. PMID 23012326